CLINICAL TRIAL: NCT04569266
Title: Effectiveness of an Exercise Re-training Program on Dyspnea in Patients After Acute Respiratory Distress Syndrome Secondary to Severe COVID-19 Pneumonia in Post-ICU
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOVER
Record Dates: First submitted 2020-09-10; First posted 2020-09-29 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-02

CONDITIONS: Dyspnea
Keywords: SARS-COV2; Pneumonia; ICU; effort re-training
MeSH Terms: conditions — Dyspnea; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No specific exercise rehabilitation treatment (Other): After randomization, patients will not benefit from any specific exercise rehabilitation treatment until 6 months post-ICU. They will then be proposed to follow the "treatment" protocol if efficacy is demonstrated, once their follow-up in the study is completed.
  Interventions: Other: No specific exercise rehabilitation treatment
- specific exercise rehabilitation treatment (Experimental): Patients will receive a prescription for exercise rehabilitation, at the rate of 2 sessions of approximately 1 hour each per week for 10 weeks.
  Continuous endurance training will start at 60-70% of the patient's maximum power. For patients who are unable to maintain continuous re-training, "interval training" sequences (30 seconds of effort followed by 30 seconds of rest) may be offered.
  Initially, the effort will be 15 minutes, then gradually increase to reach an exercise duration of 40 minutes or 45-60 minutes for endurance or interval training respectively.
  The power can be adjusted as the patient progresses to reach the target heart rate and dyspnea at 4-6 on the BORG scale.
  All patients will be offered lower limb and upper limb strengthening exercises. Each exercise will consist of 3-4 sets of 6-12 repetitions.
  Interventions: Other: Specific exercise rehabilitation treatment

INTERVENTIONS:
Other: Specific exercise rehabilitation treatment — Patients meeting the eligibility criteria will be selected consecutively. They will be contacted by telephone after at least 3 months post-resuscitation. The mMRC score is then evaluated. In case of mMRC>1, the study will then be proposed by the physiotherapist or the referring investigating physician of each participating center during this call. The patient is then offered an appointment on the reference rehabilitation platform of each center. The CDM measurement as well as the quality of life by the SF-12 scale are also carried out.
  Randomization will be stratified on the type of management during the resuscitation stay (invasive mechanical ventilation/high-flow nasal oxygen therapy) to ensure a good distribution between the 2 study arms ("control" or "treatment").
  Arms: specific exercise rehabilitation treatment
Other: No specific exercise rehabilitation treatment — Patients meeting the eligibility criteria will be selected consecutively. They will be contacted by telephone after at least 3 months post-resuscitation. The mMRC score is then evaluated. In case of mMRC>1, the study will then be proposed by the physiotherapist or the referring investigating physician of each participating center during this call. The patient is then offered an appointment on the reference rehabilitation platform of each center. The CDM measurement as well as the quality of life by the SF-12 scale are also carried out.
  Randomization will be stratified on the type of management during the resuscitation stay (invasive mechanical ventilation/high-flow nasal oxygen therapy) to ensure a good distribution between the 2 study arms ("control" or "treatment").
  Arms: No specific exercise rehabilitation treatment

SUMMARY:
Dyspnea is defined by a subjective sensation of respiratory discomfort, the intensity of which varies according to the terrain, the anamnesis and the cause. Resuscitation is associated with many causes of dyspnea, including initial distress, mechanical ventilation, or after-effects following the pathology and its management.

Respiratory distress is the most severe form of impaired lung function. It is the first cause of hospitalization in intensive care. This distress, indicative of the failure of the respiratory system, is always severe and potentially fatal. It therefore constitutes an absolute therapeutic emergency. Dyspnea is often the revealing symptom of the condition and the urgency surrounding its management is an additional factor of concern for the patient. As a result, dyspnea is a pejorative element associated with severity or even death.

DETAILED DESCRIPTION:
During these episodes of respiratory insufficiency, the management is based on ventilatory replacement by generally invasive mechanical ventilation. This allows correction of hematosis disorders but can lead to complications either directly (respiratory infections) or indirectly (neuromuscular complications and/or complications related to prolonged bed rest requiring prolonged re-education). Although mechanical ventilation makes it possible to improve the objective parameters and contributes considerably to improving the prognosis of these patients, it is nevertheless, despite the progress made, often associated with patient breathlessness due to respiratory pathology and difficulties in optimizing the interaction between the individual and the machine.

Resuscitation will also be associated with amyotrophy due to bed rest, inflammation, reduced metabolic possibilities, especially anabolic ones, and the use of certain treatments (corticosteroids, curares). This muscle loss rapidly affects the diaphragm, then secondarily the peripheral muscles in the context of resuscitation neuromyopathy. On the other hand, complications affecting the entire musculoskeletal system will quickly cause the resuscitation patient to suffer from cardiorespiratory desadaptation, reducing the capacity for exertion on discharge and ultimately resulting in dyspnea on exertion.

In patients surviving the initial condition, dyspnea persists and may be reoccurring months or even years later, despite initial rehabilitation. It is strongly associated with anxiety and even fear of death and contributes to the development of post-traumatic stress disorder. This persistent feeling of respiratory discomfort, which limits the patient's autonomy in his or her daily activities, seems to be able to reduce quality of life. Moreover, the perpetuation of this dyspnea could promote a spiral of deconditioning leading to a progressive deterioration of the cardio-respiratory system, justifying new hospitalizations.

In patients with chronic respiratory insufficiency, exercise rehabilitation supervised by physiotherapists allows, in addition to improving autonomy, a significant reduction in dyspnea, thus increasing the quality of life of these patients.

The study's objective is to evaluate the effect of post-resuscitation respiratory rehabilitation for SARS-Cov-2 in improving dyspnea. Secondly, investigators will seek to evaluate the correlation between quality of life and post-resuscitation dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years old
* Patient who has been hospitalized in an intensive care unit and discharged for at least 3 months.
* Patient who has had a laboratory confirmed respiratory infection with SARS-Cov-2 biologically confirmed by PCR or any other commercial or public health test or diagnosed by CT scan.
* Patient who has been undergoing invasive mechanical ventilation or high-flow nasal oxygen therapy during the resuscitation stay for more than 48 consecutive hours
* Francophone Patient
* Patient affiliated to social security or, failing that, to another health insurance system
* Patient capable of giving free, informed and express consent.

Exclusion Criteria:

* Lack of possibility of carrying out rehabilitation sessions :

  * Presence of contraindications to rehabilitation :

    * Severe neurological disease (Parkinson's disease, dementia, amyotrophic lateral sclerosis, aphasia, constituted ischemic stroke with significant sequelae)
    * Osteoarticular pathology reducing mobility
  * Geographic distance (>5km from the rehabilitation center's reference practice)
* Patient with a mMRC≤1
* Patient deprived of liberty
* Patient under guardianship or curatorship
* Patient under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of exercise rehabilitation on post-ICU dyspnea | Month 3
  This outcome corresponds to the comparison of Multidimensional Dyspnea Profile (MDP) scale assessment of dyspnea between month 3 and Day 1.

SECONDARY OUTCOMES:
Evaluate the effect of exercise rehabilitation on functional dyspnea | Month 3
  This outcome corresponds to the comparison of dyspnea on the Modified Medical Research Council (mMRC) scale between month 3 and day1.
Evaluate the effect of stress rehabilitation on quality of life at the end of exercise rehabilitation | Month 3
  This outcome corresponds to the comparison of Short-Form Quality of Life Assessment (SF-12) at the end of exercise rehabilitation (Month 3 by comparison day 1).

CONTACTS AND LOCATIONS:
Overall Officials: ROMANET Christophe, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (3):
- France (3):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region

REFERENCES:
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Bailey PH. The dyspnea-anxiety-dyspnea cycle--COPD patients' stories of breathlessness: "It's scary /when you can't breathe". Qual Health Res. 2004 Jul;14(6):760-78. doi: 10.1177/1049732304265973. PMID 15200799
- [Background] Ek K, Andershed B, Sahlberg-Blom E, Ternestedt BM. "The unpredictable death"-The last year of life for patients with advanced COPD: Relatives' stories. Palliat Support Care. 2015 Oct;13(5):1213-22. doi: 10.1017/S1478951514001151. Epub 2014 Oct 15. PMID 25315360
- [Background] Davidson AC; British Thoracic Society Guideline Group For The Ventilatory Management of Acute Hypercapnic Respiratory Failure in Adults. Managing acute hypercapnic respiratory failure in adults: where do we need to get to? Thorax. 2016 Apr;71(4):297-8. doi: 10.1136/thoraxjnl-2016-208281. No abstract available. PMID 26976556
- [Background] Erratum: 'British Thoracic Society Guideline Group For The Ventilatory Management of Acute Hypercapnic Respiratory Failure in Adults. Managing acute hypercapnic respiratory failure in adults: where do we need to get to?'. Thorax. 2016 Jun;71(6):492. doi: 10.1136/thoraxjnl-2016-208281corr1. No abstract available. PMID 27178824
- [Background] Howell MD, Davis AM. Management of ARDS in Adults. JAMA. 2018 Feb 20;319(7):711-712. doi: 10.1001/jama.2018.0307. No abstract available. PMID 29466577
- [Background] Gloeckl R, Marinov B, Pitta F. Practical recommendations for exercise training in patients with COPD. Eur Respir Rev. 2013 Jun 1;22(128):178-86. doi: 10.1183/09059180.00000513. PMID 23728873
- [Background] Lacasse Y, Martin S, Lasserson TJ, Goldstein RS. Meta-analysis of respiratory rehabilitation in chronic obstructive pulmonary disease. A Cochrane systematic review. Eura Medicophys. 2007 Dec;43(4):475-85. PMID 18084170
- [Background] Schmidt M, Banzett RB, Raux M, Morelot-Panzini C, Dangers L, Similowski T, Demoule A. Unrecognized suffering in the ICU: addressing dyspnea in mechanically ventilated patients. Intensive Care Med. 2014 Jan;40(1):1-10. doi: 10.1007/s00134-013-3117-3. Epub 2013 Oct 17. PMID 24132382
- [Background] Rose L, Nonoyama M, Rezaie S, Fraser I. Psychological wellbeing, health related quality of life and memories of intensive care and a specialised weaning centre reported by survivors of prolonged mechanical ventilation. Intensive Crit Care Nurs. 2014 Jun;30(3):145-51. doi: 10.1016/j.iccn.2013.11.002. Epub 2013 Dec 3. PMID 24308899
- [Background] Hough CL, Steinberg KP, Taylor Thompson B, Rubenfeld GD, Hudson LD. Intensive care unit-acquired neuromyopathy and corticosteroids in survivors of persistent ARDS. Intensive Care Med. 2009 Jan;35(1):63-8. doi: 10.1007/s00134-008-1304-4. Epub 2008 Oct 23. PMID 18946661
- [Background] Kramer CL. Intensive Care Unit-Acquired Weakness. Neurol Clin. 2017 Nov;35(4):723-736. doi: 10.1016/j.ncl.2017.06.008. PMID 28962810
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Schmidt M, Demoule A, Polito A, Porchet R, Aboab J, Siami S, Morelot-Panzini C, Similowski T, Sharshar T. Dyspnea in mechanically ventilated critically ill patients. Crit Care Med. 2011 Sep;39(9):2059-65. doi: 10.1097/CCM.0b013e31821e8779. PMID 21572329
- [Background] Binks AP, Desjardin S, Riker R. ICU Clinicians Underestimate Breathing Discomfort in Ventilated Subjects. Respir Care. 2017 Feb;62(2):150-155. doi: 10.4187/respcare.04927. Epub 2016 Dec 13. PMID 27965421
- [Result] Romanet C, Wormser J, Fels A, Lucas P, Prudat C, Sacco E, Bruel C, Plantefeve G, Pene F, Chatellier G, Philippart F. Effectiveness of exercise training on the dyspnoea of individuals with long COVID: A randomised controlled multicentre trial. Ann Phys Rehabil Med. 2023 Jun;66(5):101765. doi: 10.1016/j.rehab.2023.101765. Epub 2023 Jun 2. PMID 37271020
- See also: 1. Dangers L, Morelot-Panzini C, Schmidt M, Demoule A. Mécanismes neurophysiologiques de la dyspnée : de la perception à la clinique. Réanimation. 2014;23(4):392-401. — https://link.springer.com/article/10.1007/s13546-014-0902-4